CLINICAL TRIAL: NCT06163833
Title: MATRIx: MesenchymAl Stromal Cells for Traumatic bRain Injury
Brief Title: Mesenchymal Stromal Cells for Traumatic Brain Injury
Acronym: MATRIx
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS San Gerardo dei Tintori (Other)
Collaborators: Istituto Di Ricerche Farmacologiche Mario Negri (Other); A.O. Ospedale Papa Giovanni XXIII (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MATRIx
Record Dates: First submitted 2023-07-26; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-11

CONDITIONS: Traumatic Brain Injury With Loss of Consciousness
Keywords: mesenchimal stromal cells; neuroprotection; neurogenesis; cell therapy; synaptic plasticity; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1-control (placebo) (Placebo Comparator): Administration: once (bolus), intravenous, 36mL
  Interventions: Other: Placebo-storage solution
- 2-MSCs 80*10^6 (Experimental): Administration: once (bolus), intravenous, 36mL
  Interventions: Drug: Mesenchymal stromal cell low dosage-80*10^6 cells
- 3-MSCs 160*10^6 (Experimental): Administration: once (bolus), intravenous, 36mL
  Interventions: Drug: Mesenchymal stromal cell low dosage-160*10^6 cells

INTERVENTIONS:
Drug: Mesenchymal stromal cell low dosage-80*10^6 cells — MSCs have to be administered at the dosage of 80*10^6. MSCs have to be administered by intravenous infusion via an in situ venous catheter within 15 minutes from the preparation and within 48 hours from TBI.
  They have to be diluted 1:2 in a saline solution for a total of 36mL.
  Other Names: MATRIx MSC low dose
  Arms: 2-MSCs 80*10^6
Drug: Mesenchymal stromal cell low dosage-160*10^6 cells — MSCs have to be administered at the dosage of 160*10^6. MSCs have to be administered by intravenous infusion via an in situ venous catheter within 15 minutes from the preparation and within 48 hours from TBI.
  They have to be diluted 1:2 in a saline solution for a total of 36mL.
  Other Names: MATRIx MSC high dose
  Arms: 3-MSCs 160*10^6
Other: Placebo-storage solution — Placebo has to be administered by intravenous infusion via an in situ venous catheter within 15 minutes from the preparation and within 48 hours from TBI. It has to be diluted 1:2 in a saline solution for a total of 36mL.
  Other Names: MATRIx placebo
  Arms: 1-control (placebo)

SUMMARY:
Traumatic Brain Injury (TBI) is an alteration of brain function caused by an external force. Long-term mortality in TBI is substantial, TBI survivors can develop chronic progressive disabilities and have a life expectancy shortened by 6 years. Treatment consists in supportive therapy directed at prevention of second insults, but no neuroprotective therapy is available. Given the multifaceted nature of TBI, mesenchymal stromal cells (MSCs) are an ideal candidate: they release multiple soluble factors shown to ameliorate the injury microenvironment through immunomodulatory, protective, reparative and regenerative processes. Preclinical data across a range of different TBI models and injury severities show that human MSCs improve outcome through pleiotropic mechanisms of protection and repair. Thus, data indicate MSCs as strong therapeutic candidate and support a clinical study in TBI.

Aim: the study is designed to assess the safety and the efficacy of the MSCs, intravenously administered in severe TBI patients within 48h from injury. The study will be conducted in a stepwise manner. Step 1 will enroll 36 patients (randomized 1:1:1 in arms 80 x 10^6 MSCs vs 160 x 10^6 MSCs vs placebo) to define safety, and will allow to select the most promising dose. Step 2 will enroll 30 patients (1:1 in arms MSCs selected dose vs placebo) to define the MSC activity based on the quantification of the plasmatic levels of the neurofilament light (NFL) at 14 days, as biomarker of neuronal damage.

Secondary objectives are aimed to assess:

1. brain injury evolution and white matter damage by longitudinal neuroimaging (at 4 days and 14 days post-TBI and at 6 months)
2. brain immunomodulatory changes by temporal profiling of circulating biomarkers of brain damage and neuroinflammation (daily for 3 days after TBI, at day 7 and 14, and at 1, 6 and 12 months)
3. clinical outcome by a structured clinical and neuropsychological assessment at both 6 and 12 months

Methods: a multicenter, double blind, randomized, placebo-controlled, adaptive phase II dose finding study.

Duration of the study: 36 months (24 of enrolment and 12 of follow up).

Funding: Fondazione Regionale per la ricerca Biomedica, FRRB (Call "Unmet medical needs", proposal number 3440227) and Italian Ministry of health (Ministero della Salute, Bando di Ricerca Finalizzata 2021; proposal number RF-2021-12372642).

DETAILED DESCRIPTION:
Study Description: Multicenter, double blind, randomized, placebo-controlled, adaptive phase II dose finding study meant to define if MSCs, administered at dosage of 80 or 160 x 10^6 cells within 48h from TBI, are safe in patients with severe TBI, and to define if MSCs, administered at the dosage found to be safe and more promising, decrease the plasmatic neurofilament light (NFL) biomarker of brain damage at 14 days. Patients will be recruited at the Neurointensive Care Unit at Fondazione IRCCS San Gerardo dei Tintori, Monza, at ASST Ospedale Papa Giovanni XXIII Bergamo and at Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico of Milano. Collection of multiple clinical, neuroimaging and biological parameters will describe TBI evolution.

Preclinical studies: Studies in rodent TBI models have shown that administration of MSCs produces functional improvement with amelioration of sensorimotor and cognitive deficit, reduction of contusion volume and neuronal loss, modulation of the inflammatory response with decreased inflammation, stimulation of beneficial endogenous mechanisms (angiogenesis, neurogenesis, synaptic plasticity). These results support the notion that MSCs can reprogram the microenvironment mitigating the progression of brain damage and fostering recovery of function. Only few clinical studies have assessed the safety, feasibility and efficacy of MSC therapy. No adverse events (AEs) or severe adverse events (SAEs) were reported. No AEs were associated to the intravenous route, which is the one the investigators propose for the study.

Target Sample Size:The total number of evaluable patients to be analyzed will be 66 (27 on the control arm, 12 in the experimental arm stopping at first step and 27 in the experimental arm reaching the second step). In details, the total number of evaluable patients to be analyzed will be 24 (12 patients in each experimental arm) for the safety interim analysis and 54 for the final efficacy analysis (27 patients in both the control arm and in the experimental arm reaching the second step).

Expecting a 13% of deaths of TBI patients in ICU, the number of patients to be randomized is about 78 (32 in the control arm, 14 in the experimental arm stopping at first step and 32 in the experimental arm reaching the second step). In case of the trial closure after the first step, the number of patients to randomize will be about 42 (14 in each arm).

Statistical design and sample size:The statistical study design is conceived in 2 steps.

Step 1: An interim safety analysis will be performed to evaluate separately in each of the two experimental dosage groups, at one-sided type I error rate of 10%, whether more than 30% of patients experience at least one serious adverse drug reaction (SADR) within 14 days from treatment, and at the same time at a power of 80% whether 5% or less of the patients do not experience any SADR. Adopting the Fleming design with A'Hern's approach, 12 evaluable patients will be analyzed in each group (36 patients overall). The maximum number of patients experiencing at least one SADR to observe in each experimental group is 1 out of 12, since this result is associated with an upper limit of the 80% exact confidence interval of 28.8%.

The experimental treatment will be considered as safe for this step only if none or one patient experiment a SADR.

According to the above role:

* if both experimental treatments are considered not safe, the study will be stopped for safety issues and the step 2 of the study will not be performed
* if one experimental treatment is considered safe and the other not safe, only the safe arm will proceed with the step 2 of the study
* if both the experimental dosages are safe, then the more active schedule will be selected for the step 2 The more active schedule will be defined in terms of proportion of patients who reaches a NFL increase at 14 days equal or lower than baseline level by 5 folds (defined as "responder patients").

This cut-off has been defined based on longitudinal quantification kindly provided by BIO-AX-TBI collaborators, showing a median increase of 12.8-fold at 14 days compared to baseline, with first quartile equal to 5-fold increase (see paragraph 5.4 for details). In case of an equal number of responder patients in the two experimental arms, the cut-off defining the response will be increased by 1 unit iteratively since a difference between the two experimental arms will be observed. This assessment will only be performed on the MSC treated arms; the control group will not be considered. According to Simon, Wittes and Ellemberg randomized phase II design, the study has more than 80% probability of correctly select the more active schedule when the proportion of responder patients is 15% higher in the first of the two schedules of treatment.

Step 2: the primary endpoint will be the NFL at 14 days. The final efficacy analysis will be performed by increasing the sample size to 27 evaluable patients in the experimental and control arms. The study is designed to detect an effect size of 0.59 on logarithmic scale of the experimental to control arm, setting a one-sided type I error rate of 10% and a power of 80%.

Data will be analysed by the study biostatistician using the software SAS 9.4 release. A full Statistical Analysis Plan will be written prior to statistical analysis.

Deceased or lost to follow-up patients and patients with missing values will contribute to the analysis of the secondary outcomes only for the time during which data are available.

All patients who have received the treatment will be included in the safety analysis. Each patient will be analyzed in the arm actually received.

The assessment of safety will be mainly based on adverse reactions (ARs) and the frequency and nature of the serious adverse events (SAEs) and will be conducted on the safety analysis set.

Expected results: the investigators expect to prove the safety and efficacy of MSC intravenous administration in acute and severe TBI patients. The investigators will provide a detailed longitudinal description of the effects of MSCs on brain advanced neuroimaging trajectories, on axonal damage and neuro-immunomodulatory changes by blood biomarker analysis and on clinical outcome.

MSC preparation: The preparation of MSCs will be performed as detailed in the IMP brochure according to Good Manufacturing Procedures (GMP) guidelines at Laboratorio Stefano Verri, ASST MONZA. Laboratorio Stefano Verri has standard operating procedures in place for storage, release, thawing, preparing and administering the MSCs.

MSCs are stored in vials containing 40 X 10^6 MSCs each in 4.5 ml of storage solution (2.5 ml albumin 20%, 1.1 ml normal saline solution, 0.45 ml citrate-dextrose solution (ACD), 0.45 ml Dimethyl sulfoxide (DMSO)). Vials containing 4.5 ml of storage solution only will be prepared and stored in the same manner. The MSC injections and the placebo injections will have identical appearance and consistency. Vials are stored in the vapor phase of liquid nitrogen until the time of administration.

The study treatment will be prepared by qualified personnel under a class A laminar flow hood in proximity to the ICU.

IMP will be administered acutely (within 48h after injury) within 15 minutes from the preparation through a central venous line.

Random allocation procedure: Patients will be randomly assigned to one of the three treatment groups (allocation ratio 1:1:1 for the first step and 1:1 for the second step). The study biostatistician will prepare the sequence of treatments according to a randomized permuted blocks procedure. The randomization schedule will be generated using SAS 9.4 release. The randomized allocation of treatment will be centralized.

Upon recruitment of a patient meeting the inclusion criteria, the local investigator will follow a randomization list (provided by the factory member's personnel) (detailed in the Manual of Procedures) to assign the treatment to the patient in a blinded fashion manner.

Blinding: The subjects, the research coordinators and investigators, and the personnel involved in outcomes assessments and monitoring compliance will all be blinded. Treatment assignment will be known only to the Sponsor Data Management Team and the Cell Factory of each center. An unblinded physician will be designated to monitor safety results.

Patient withdrawal: Patients may withdraw (or be withdrawn) from the study at any time. Withdrawals within 14 days will be replaced.

Reasons for patient withdrawal include:

* Adverse event that in the judgement of the Investigator requires study withdrawal
* Patient wishes to withdraw from the study
* Patient is lost to follow-up Benefit/Risk assessment: The use of MSC therapy for TBI patients is experimental and may not result in any direct benefit to the patient. Nevertheless, proposers strongly believe that the benefits awaited from this MSC-based therapeutic strategy is an amelioration of the evolution of TBI pathology with a consequent better outcome with the reduction of the long-term disabilities. MSCs are a particularly promising cell therapy because of their availability, immunologic properties and track record of safety and efficacy.

The risks associated with the intravenous administration procedure include bleeding, swelling and minor pain on injection. These are self-limiting and do not pose any long-term problem.

During the first few hours from the MSC intravenous infusion: headache, fever, rush and allergic reaction may appear. The risk of allergic reaction is mitigated by the use of human platelet lysate instead of the fetal calf serum during the manufacturing process. This also allows to avoid the possible transmission of still unknown zoonosis.

There is also a remote infectious risk that can be treated with appropriate antibiotics. The infection may conduct pain, discomfort and tissue damage.

A possible risk of intravenous MSC infusion is represented by thromboembolic events. MSC infusion could increase pulmonary vascular resistance in the presence of injured pulmonary microcirculation, potentially by aggregating or clumping in capillaries or small arterioles. Subsequent potential risks are acute right heart failure, impaired cardiac output and hemodynamic instability. Additionally, infusion of MSCs could potentially worsen ventilation-perfusion mismatch and result in further impairment of oxygenation or carbon dioxide excretion.

Collection of Data: All data obtained during this clinical trial will be captured electronically in a project specific programmed Electronic Data Capture (EDC) application.

For each subject, all data and trial-related visits will be recorded in the eCRF (electronic Case Report Form). If a subject withdraws from the trial, the reason must be stated in the eCRF.

Informed consent: It is the responsibility of the investigator/delegate to obtain informed consent according to ICH-GCP and Declaration of Helsinki guidelines and local regulations from each individual subject participating in this study and/or his/her legally designated representative/proxy. If the subject is not able to provide personal consent at the time the consent is obtained, then he/she must provide or withdraw this consent as soon as possible once his/her clinical condition has improved to the extent that providing personal consent is possible, unless local regulations state otherwise.

The informed consent form (ICF) will be provided in the country's local language(s).

Regulatory and Ethical Compliance: The trial will be performed in accordance with the Declaration of Helsinki and the Good Clinical Practice. The trial obtained the Regulatory Agency (AIFA) approval. The protocol and trial conduct will comply with the Medicines for Human Use (Clinical Trials) Regulations 2004 and any relevant amendments. Development Safety Update Reports will be submitted to the IEC and Regulatory Agency.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years
* Clinical frailty index (CFI) < 5
* Evidence of TBI confirmed by abnormalities consistent with trauma on CT scan upon admission (Marshall's CT Classification >1)
* Feasibility of study drug (MSC/placebo) administration within 48 hours from TBI
* GCS ≤ 8 at recruitment and at least one pupil reactive to light
* ICP monitoring already inserted or planned for clinical indications
* Weight < 100 Kg and > 40 kg

Exclusion Criteria:

* Motor GCS > 5 at recruitment
* High likelihood (> 85%) of death in the first 48 h calculated by IMPACT calculator on early admission data
* Bilateral mydriasis
* Opening ICP > 40 mmHg
* Known history of prior brain injury, psychiatric disorder, neurological impairment and/or deficit
* Brain penetrating injury
* Spinal cord injury
* Previous epilepsy requiring anti-convulsant therapy
* Severe organ failure (including PaO2/FiO2<200 and shock)
* Recent serious infectious process
* Cancer
* Immunosuppression
* Human immunodeficiency virus
* Positive urine pregnancy test or nursing
* Known risk/history of coagulopathy and thromboembolism
* Pre-existing and severe:

  * lung disease (such as asthma, chronic obstructive pulmonary disease),
  * heart dysfunction (as heart failure and reduced cardiac output),
  * liver insufficiency (as cirrhosis)
  * kidney insufficiency
  * and other organ severe abnormalities
* Known hypersensitivity to excipients used in the formulation (Dimethyl sulfoxide (DMSO), Citrate-dextrose solution (ACD))
* Participation in a concurrent interventional study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
safety of mesenchimal stromal cell intravenous administration in TBI patients | 14 days from treatment administration
  number of patients in each of the two experimental dosage group experiencing at least one serious adverse drug reaction (SADR) (assessed by CTCAE v5.0) within 14 days from treatment. The maximum number of patients experiencing at least one SADR to observe in each experimental group is 1 out of 12.
efficacy of mesenchimal stromal cells in preventing subacutely post-TBI brain axonal injury | 14 days post-TBI
  number of MSC-treated patients who reach a plasmatic NFL (neurofilament light) increase at 14 days post-treatment equal or lower than 5-fold compared to the baseline (these patients are defined as "responder patients")

SECONDARY OUTCOMES:
efficacy of mesenchimal stromal cells in preventing post-TBI brain anatomical injury | 4 days post-TBI, 14 days and 6 months
  number of MSC-treated patients that show an improvement in terms of atrophy, diffusion and myelin integrity detected by longitudinal advanced MRI performed acutely (at 4 days post-TBI), subacutely (at 14 days) and at 6 months post-TBI.
efficacy of mesenchimal stromal cells in preventing the plasmatic increase of TBI-related circulating biomarkers | daily for 3 days after TBI, at day 7 and 14, and at 1, 6 and 12 months
  number of patients who have decreased values of markers related to axonal damage (NFL, GFAP), neuroinflammation (IL-6, IL-10, TNFa) and vascular damage (MMP9) evaluated daily for 3 days after TBI, at day 7 and 14, and at 1, 6 and 12 months
efficacy of mesenchimal stromal cell administration in improving the clinical outcome of TBI patients | 6 and 12 months post-TBI
  number of patients with an improved clinical and neuropsychological outcome at both 6 and 12 months evaluated by the administration of structured clinical and neuropsychological questionnaires (Glasgow Outcome Scale Extended (GOSE) and quality of life after brain injury test (QOLIBRI)).

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Citerio, Professor, Principal Investigator — Fondazione IRCCS San Gerardo dei Tintori
Locations (3):
- Italy (3):
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, MB
  - ASST Ospedale Papa Giovanni XXIII Bergamo, Bergamo
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico of Milano, Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ng SY, Lee AYW. Traumatic Brain Injuries: Pathophysiology and Potential Therapeutic Targets. Front Cell Neurosci. 2019 Nov 27;13:528. doi: 10.3389/fncel.2019.00528. eCollection 2019. PMID 31827423
- [Background] Steyerberg EW, Wiegers E, Sewalt C, Buki A, Citerio G, De Keyser V, Ercole A, Kunzmann K, Lanyon L, Lecky F, Lingsma H, Manley G, Nelson D, Peul W, Stocchetti N, von Steinbuchel N, Vande Vyvere T, Verheyden J, Wilson L, Maas AIR, Menon DK; CENTER-TBI Participants and Investigators. Case-mix, care pathways, and outcomes in patients with traumatic brain injury in CENTER-TBI: a European prospective, multicentre, longitudinal, cohort study. Lancet Neurol. 2019 Oct;18(10):923-934. doi: 10.1016/S1474-4422(19)30232-7. PMID 31526754
- [Background] Voormolen DC, Polinder S, von Steinbuechel N, Feng Y, Wilson L, Oppe M, Haagsma JA; CENTER-TBI participants and investigators. Health-related quality of life after traumatic brain injury: deriving value sets for the QOLIBRI-OS for Italy, The Netherlands and The United Kingdom. Qual Life Res. 2020 Nov;29(11):3095-3107. doi: 10.1007/s11136-020-02583-6. Epub 2020 Jul 15. PMID 32671617
- [Background] Maas AIR, Menon DK, Adelson PD, Andelic N, Bell MJ, Belli A, Bragge P, Brazinova A, Buki A, Chesnut RM, Citerio G, Coburn M, Cooper DJ, Crowder AT, Czeiter E, Czosnyka M, Diaz-Arrastia R, Dreier JP, Duhaime AC, Ercole A, van Essen TA, Feigin VL, Gao G, Giacino J, Gonzalez-Lara LE, Gruen RL, Gupta D, Hartings JA, Hill S, Jiang JY, Ketharanathan N, Kompanje EJO, Lanyon L, Laureys S, Lecky F, Levin H, Lingsma HF, Maegele M, Majdan M, Manley G, Marsteller J, Mascia L, McFadyen C, Mondello S, Newcombe V, Palotie A, Parizel PM, Peul W, Piercy J, Polinder S, Puybasset L, Rasmussen TE, Rossaint R, Smielewski P, Soderberg J, Stanworth SJ, Stein MB, von Steinbuchel N, Stewart W, Steyerberg EW, Stocchetti N, Synnot A, Te Ao B, Tenovuo O, Theadom A, Tibboel D, Videtta W, Wang KKW, Williams WH, Wilson L, Yaffe K; InTBIR Participants and Investigators. Traumatic brain injury: integrated approaches to improve prevention, clinical care, and research. Lancet Neurol. 2017 Dec;16(12):987-1048. doi: 10.1016/S1474-4422(17)30371-X. Epub 2017 Nov 6. No abstract available. PMID 29122524
- [Background] Carbonara M, Fossi F, Zoerle T, Ortolano F, Moro F, Pischiutta F, Zanier ER, Stocchetti N. Neuroprotection in Traumatic Brain Injury: Mesenchymal Stromal Cells can Potentially Overcome Some Limitations of Previous Clinical Trials. Front Neurol. 2018 Oct 24;9:885. doi: 10.3389/fneur.2018.00885. eCollection 2018. PMID 30405517
- [Background] Cossu G, Birchall M, Brown T, De Coppi P, Culme-Seymour E, Gibbon S, Hitchcock J, Mason C, Montgomery J, Morris S, Muntoni F, Napier D, Owji N, Prasad A, Round J, Saprai P, Stilgoe J, Thrasher A, Wilson J. Lancet Commission: Stem cells and regenerative medicine. Lancet. 2018 Mar 3;391(10123):883-910. doi: 10.1016/S0140-6736(17)31366-1. Epub 2017 Oct 4. No abstract available. PMID 28987452
- [Background] Fu Y, Karbaat L, Wu L, Leijten J, Both SK, Karperien M. Trophic Effects of Mesenchymal Stem Cells in Tissue Regeneration. Tissue Eng Part B Rev. 2017 Dec;23(6):515-528. doi: 10.1089/ten.TEB.2016.0365. PMID 28490258
- [Background] Lin CH, Lin W, Su YC, Cheng-Yo Hsuan Y, Chen YC, Chang CP, Chou W, Lin KC. Modulation of parietal cytokine and chemokine gene profiles by mesenchymal stem cell as a basis for neurotrauma recovery. J Formos Med Assoc. 2019 Dec;118(12):1661-1673. doi: 10.1016/j.jfma.2019.01.008. Epub 2019 Jan 30. PMID 30709695
- [Background] Zanier ER, Montinaro M, Vigano M, Villa P, Fumagalli S, Pischiutta F, Longhi L, Leoni ML, Rebulla P, Stocchetti N, Lazzari L, De Simoni MG. Human umbilical cord blood mesenchymal stem cells protect mice brain after trauma. Crit Care Med. 2011 Nov;39(11):2501-10. doi: 10.1097/CCM.0b013e31822629ba. PMID 21725237
- [Background] Zanier ER, Pischiutta F, Riganti L, Marchesi F, Turola E, Fumagalli S, Perego C, Parotto E, Vinci P, Veglianese P, D'Amico G, Verderio C, De Simoni MG. Bone marrow mesenchymal stromal cells drive protective M2 microglia polarization after brain trauma. Neurotherapeutics. 2014 Jul;11(3):679-95. doi: 10.1007/s13311-014-0277-y. PMID 24965140
- [Background] Pischiutta F, D'Amico G, Dander E, Biondi A, Biagi E, Citerio G, De Simoni MG, Zanier ER. Immunosuppression does not affect human bone marrow mesenchymal stromal cell efficacy after transplantation in traumatized mice brain. Neuropharmacology. 2014 Apr;79:119-26. doi: 10.1016/j.neuropharm.2013.11.001. Epub 2013 Nov 15. PMID 24246661
- [Background] Pischiutta F, Brunelli L, Romele P, Silini A, Sammali E, Paracchini L, Marchini S, Talamini L, Bigini P, Boncoraglio GB, Pastorelli R, De Simoni MG, Parolini O, Zanier ER. Protection of Brain Injury by Amniotic Mesenchymal Stromal Cell-Secreted Metabolites. Crit Care Med. 2016 Nov;44(11):e1118-e1131. doi: 10.1097/CCM.0000000000001864. PMID 27441900
- [Background] Lalu MM, McIntyre L, Pugliese C, Fergusson D, Winston BW, Marshall JC, Granton J, Stewart DJ; Canadian Critical Care Trials Group. Safety of cell therapy with mesenchymal stromal cells (SafeCell): a systematic review and meta-analysis of clinical trials. PLoS One. 2012;7(10):e47559. doi: 10.1371/journal.pone.0047559. Epub 2012 Oct 25. PMID 23133515
- [Background] Diez-Tejedor E, Gutierrez-Fernandez M, Martinez-Sanchez P, Rodriguez-Frutos B, Ruiz-Ares G, Lara ML, Gimeno BF. Reparative therapy for acute ischemic stroke with allogeneic mesenchymal stem cells from adipose tissue: a safety assessment: a phase II randomized, double-blind, placebo-controlled, single-center, pilot clinical trial. J Stroke Cerebrovasc Dis. 2014 Nov-Dec;23(10):2694-2700. doi: 10.1016/j.jstrokecerebrovasdis.2014.06.011. Epub 2014 Oct 7. PMID 25304723
- [Background] Levy ML, Crawford JR, Dib N, Verkh L, Tankovich N, Cramer SC. Phase I/II Study of Safety and Preliminary Efficacy of Intravenous Allogeneic Mesenchymal Stem Cells in Chronic Stroke. Stroke. 2019 Oct;50(10):2835-2841. doi: 10.1161/STROKEAHA.119.026318. Epub 2019 Sep 9. PMID 31495331
- [Background] Care AD, Ross R. Fetal calcium homeostasis. J Dev Physiol. 1984 Feb;6(1):59-66. No abstract available. PMID 6423725
- [Background] Dewan MC, Rattani A, Gupta S, Baticulon RE, Hung YC, Punchak M, Agrawal A, Adeleye AO, Shrime MG, Rubiano AM, Rosenfeld JV, Park KB. Estimating the global incidence of traumatic brain injury. J Neurosurg. 2018 Apr 27;130(4):1080-1097. doi: 10.3171/2017.10.JNS17352. Print 2019 Apr 1. PMID 29701556
- [Background] Majdan M, Plancikova D, Brazinova A, Rusnak M, Nieboer D, Feigin V, Maas A. Epidemiology of traumatic brain injuries in Europe: a cross-sectional analysis. Lancet Public Health. 2016 Dec;1(2):e76-e83. doi: 10.1016/S2468-2667(16)30017-2. Epub 2016 Nov 29. PMID 29253420
- [Background] Stocchetti N, Zanier ER. Chronic impact of traumatic brain injury on outcome and quality of life: a narrative review. Crit Care. 2016 Jun 21;20(1):148. doi: 10.1186/s13054-016-1318-1. PMID 27323708
- [Background] Blennow K, Brody DL, Kochanek PM, Levin H, McKee A, Ribbers GM, Yaffe K, Zetterberg H. Traumatic brain injuries. Nat Rev Dis Primers. 2016 Nov 17;2:16084. doi: 10.1038/nrdp.2016.84. PMID 27853132
- [Background] Das M, Mayilsamy K, Mohapatra SS, Mohapatra S. Mesenchymal stem cell therapy for the treatment of traumatic brain injury: progress and prospects. Rev Neurosci. 2019 Nov 26;30(8):839-855. doi: 10.1515/revneuro-2019-0002. PMID 31203262
- [Background] Roberts I, Yates D, Sandercock P, Farrell B, Wasserberg J, Lomas G, Cottingham R, Svoboda P, Brayley N, Mazairac G, Laloe V, Munoz-Sanchez A, Arango M, Hartzenberg B, Khamis H, Yutthakasemsunt S, Komolafe E, Olldashi F, Yadav Y, Murillo-Cabezas F, Shakur H, Edwards P; CRASH trial collaborators. Effect of intravenous corticosteroids on death within 14 days in 10008 adults with clinically significant head injury (MRC CRASH trial): randomised placebo-controlled trial. Lancet. 2004 Oct 9-15;364(9442):1321-8. doi: 10.1016/S0140-6736(04)17188-2. PMID 15474134
- [Background] Temkin NR, Anderson GD, Winn HR, Ellenbogen RG, Britz GW, Schuster J, Lucas T, Newell DW, Mansfield PN, Machamer JE, Barber J, Dikmen SS. Magnesium sulfate for neuroprotection after traumatic brain injury: a randomised controlled trial. Lancet Neurol. 2007 Jan;6(1):29-38. doi: 10.1016/S1474-4422(06)70630-5. PMID 17166799
- [Background] Wright DW, Yeatts SD, Silbergleit R, Palesch YY, Hertzberg VS, Frankel M, Goldstein FC, Caveney AF, Howlett-Smith H, Bengelink EM, Manley GT, Merck LH, Janis LS, Barsan WG; NETT Investigators. Very early administration of progesterone for acute traumatic brain injury. N Engl J Med. 2014 Dec 25;371(26):2457-66. doi: 10.1056/NEJMoa1404304. Epub 2014 Dec 10. PMID 25493974
- [Background] Diaz-Arrastia R, Kochanek PM, Bergold P, Kenney K, Marx CE, Grimes CJ, Loh LT, Adam LT, Oskvig D, Curley KC, Salzer W. Pharmacotherapy of traumatic brain injury: state of the science and the road forward: report of the Department of Defense Neurotrauma Pharmacology Workgroup. J Neurotrauma. 2014 Jan 15;31(2):135-58. doi: 10.1089/neu.2013.3019. PMID 23968241
- [Background] Edwards P, Arango M, Balica L, Cottingham R, El-Sayed H, Farrell B, Fernandes J, Gogichaisvili T, Golden N, Hartzenberg B, Husain M, Ulloa MI, Jerbi Z, Khamis H, Komolafe E, Laloe V, Lomas G, Ludwig S, Mazairac G, Munoz Sanchez Mde L, Nasi L, Olldashi F, Plunkett P, Roberts I, Sandercock P, Shakur H, Soler C, Stocker R, Svoboda P, Trenkler S, Venkataramana NK, Wasserberg J, Yates D, Yutthakasemsunt S; CRASH trial collaborators. Final results of MRC CRASH, a randomised placebo-controlled trial of intravenous corticosteroid in adults with head injury-outcomes at 6 months. Lancet. 2005 Jun 4-10;365(9475):1957-9. doi: 10.1016/S0140-6736(05)66552-X. PMID 15936423
- [Background] Zafonte RD, Bagiella E, Ansel BM, Novack TA, Friedewald WT, Hesdorffer DC, Timmons SD, Jallo J, Eisenberg H, Hart T, Ricker JH, Diaz-Arrastia R, Merchant RE, Temkin NR, Melton S, Dikmen SS. Effect of citicoline on functional and cognitive status among patients with traumatic brain injury: Citicoline Brain Injury Treatment Trial (COBRIT). JAMA. 2012 Nov 21;308(19):1993-2000. doi: 10.1001/jama.2012.13256. PMID 23168823
- [Background] Skolnick BE, Maas AI, Narayan RK, van der Hoop RG, MacAllister T, Ward JD, Nelson NR, Stocchetti N; SYNAPSE Trial Investigators. A clinical trial of progesterone for severe traumatic brain injury. N Engl J Med. 2014 Dec 25;371(26):2467-76. doi: 10.1056/NEJMoa1411090. Epub 2014 Dec 10. PMID 25493978
- [Background] Cooper DJ, Nichol AD, Bailey M, Bernard S, Cameron PA, Pili-Floury S, Forbes A, Gantner D, Higgins AM, Huet O, Kasza J, Murray L, Newby L, Presneill JJ, Rashford S, Rosenfeld JV, Stephenson M, Vallance S, Varma D, Webb SAR, Trapani T, McArthur C; POLAR Trial Investigators and the ANZICS Clinical Trials Group. Effect of Early Sustained Prophylactic Hypothermia on Neurologic Outcomes Among Patients With Severe Traumatic Brain Injury: The POLAR Randomized Clinical Trial. JAMA. 2018 Dec 4;320(21):2211-2220. doi: 10.1001/jama.2018.17075. PMID 30357266
- [Background] Wilson L, Stewart W, Dams-O'Connor K, Diaz-Arrastia R, Horton L, Menon DK, Polinder S. The chronic and evolving neurological consequences of traumatic brain injury. Lancet Neurol. 2017 Oct;16(10):813-825. doi: 10.1016/S1474-4422(17)30279-X. Epub 2017 Sep 12. PMID 28920887
- [Background] Friedenstein AJ, Chailakhjan RK, Lalykina KS. The development of fibroblast colonies in monolayer cultures of guinea-pig bone marrow and spleen cells. Cell Tissue Kinet. 1970 Oct;3(4):393-403. doi: 10.1111/j.1365-2184.1970.tb00347.x. No abstract available. PMID 5523063
- [Background] Karp JM, Leng Teo GS. Mesenchymal stem cell homing: the devil is in the details. Cell Stem Cell. 2009 Mar 6;4(3):206-16. doi: 10.1016/j.stem.2009.02.001. PMID 19265660
- [Background] Li Y, Chen J, Chen XG, Wang L, Gautam SC, Xu YX, Katakowski M, Zhang LJ, Lu M, Janakiraman N, Chopp M. Human marrow stromal cell therapy for stroke in rat: neurotrophins and functional recovery. Neurology. 2002 Aug 27;59(4):514-23. doi: 10.1212/wnl.59.4.514. PMID 12196642
- [Background] Li J, Zhu H, Liu Y, Li Q, Lu S, Feng M, Xu Y, Huang L, Ma C, An Y, Zhao RC, Wang R, Qin C. Human mesenchymal stem cell transplantation protects against cerebral ischemic injury and upregulates interleukin-10 expression in Macacafascicularis. Brain Res. 2010 Jun 2;1334:65-72. doi: 10.1016/j.brainres.2010.03.080. Epub 2010 Mar 28. PMID 20353760
- [Background] Xin H, Li Y, Shen LH, Liu X, Wang X, Zhang J, Pourabdollah-Nejad D S, Zhang C, Zhang L, Jiang H, Zhang ZG, Chopp M. Increasing tPA activity in astrocytes induced by multipotent mesenchymal stromal cells facilitate neurite outgrowth after stroke in the mouse. PLoS One. 2010 Feb 3;5(2):e9027. doi: 10.1371/journal.pone.0009027. PMID 20140248
- [Background] Ohtaki H, Ylostalo JH, Foraker JE, Robinson AP, Reger RL, Shioda S, Prockop DJ. Stem/progenitor cells from bone marrow decrease neuronal death in global ischemia by modulation of inflammatory/immune responses. Proc Natl Acad Sci U S A. 2008 Sep 23;105(38):14638-43. doi: 10.1073/pnas.0803670105. Epub 2008 Sep 15. PMID 18794523
- [Background] Zhang R, Liu Y, Yan K, Chen L, Chen XR, Li P, Chen FF, Jiang XD. Anti-inflammatory and immunomodulatory mechanisms of mesenchymal stem cell transplantation in experimental traumatic brain injury. J Neuroinflammation. 2013 Aug 23;10:106. doi: 10.1186/1742-2094-10-106. PMID 23971414
- [Background] Peruzzaro ST, Andrews MMM, Al-Gharaibeh A, Pupiec O, Resk M, Story D, Maiti P, Rossignol J, Dunbar GL. Transplantation of mesenchymal stem cells genetically engineered to overexpress interleukin-10 promotes alternative inflammatory response in rat model of traumatic brain injury. J Neuroinflammation. 2019 Jan 5;16(1):2. doi: 10.1186/s12974-018-1383-2. PMID 30611291
- [Background] Pischiutta F, Caruso E, Cavaleiro H, Salgado AJ, Loane DJ, Zanier ER. Mesenchymal stromal cell secretome for traumatic brain injury: Focus on immunomodulatory action. Exp Neurol. 2022 Nov;357:114199. doi: 10.1016/j.expneurol.2022.114199. Epub 2022 Aug 8. PMID 35952763
- [Background] Menge T, Zhao Y, Zhao J, Wataha K, Gerber M, Zhang J, Letourneau P, Redell J, Shen L, Wang J, Peng Z, Xue H, Kozar R, Cox CS Jr, Khakoo AY, Holcomb JB, Dash PK, Pati S. Mesenchymal stem cells regulate blood-brain barrier integrity through TIMP3 release after traumatic brain injury. Sci Transl Med. 2012 Nov 21;4(161):161ra150. doi: 10.1126/scitranslmed.3004660. PMID 23175708
- [Background] Zacharek A, Chen J, Cui X, Li A, Li Y, Roberts C, Feng Y, Gao Q, Chopp M. Angiopoietin1/Tie2 and VEGF/Flk1 induced by MSC treatment amplifies angiogenesis and vascular stabilization after stroke. J Cereb Blood Flow Metab. 2007 Oct;27(10):1684-91. doi: 10.1038/sj.jcbfm.9600475. Epub 2007 Mar 14. PMID 17356562
- [Background] Yoo SW, Kim SS, Lee SY, Lee HS, Kim HS, Lee YD, Suh-Kim H. Mesenchymal stem cells promote proliferation of endogenous neural stem cells and survival of newborn cells in a rat stroke model. Exp Mol Med. 2008 Aug 31;40(4):387-97. doi: 10.3858/emm.2008.40.4.387. PMID 18779651
- [Background] Bao X, Wei J, Feng M, Lu S, Li G, Dou W, Ma W, Ma S, An Y, Qin C, Zhao RC, Wang R. Transplantation of human bone marrow-derived mesenchymal stem cells promotes behavioral recovery and endogenous neurogenesis after cerebral ischemia in rats. Brain Res. 2011 Jan 7;1367:103-13. doi: 10.1016/j.brainres.2010.10.063. Epub 2010 Oct 23. PMID 20977892
- [Background] Gutierrez-Fernandez M, Rodriguez-Frutos B, Ramos-Cejudo J, Teresa Vallejo-Cremades M, Fuentes B, Cerdan S, Diez-Tejedor E. Effects of intravenous administration of allogenic bone marrow- and adipose tissue-derived mesenchymal stem cells on functional recovery and brain repair markers in experimental ischemic stroke. Stem Cell Res Ther. 2013 Jan 28;4(1):11. doi: 10.1186/scrt159. PMID 23356495
- [Background] Lu D, Mahmood A, Wang L, Li Y, Lu M, Chopp M. Adult bone marrow stromal cells administered intravenously to rats after traumatic brain injury migrate into brain and improve neurological outcome. Neuroreport. 2001 Mar 5;12(3):559-63. doi: 10.1097/00001756-200103050-00025. PMID 11234763
- [Background] Gennai S, Monsel A, Hao Q, Liu J, Gudapati V, Barbier EL, Lee JW. Cell-based therapy for traumatic brain injury. Br J Anaesth. 2015 Aug;115(2):203-12. doi: 10.1093/bja/aev229. PMID 26170348
- [Background] Peng W, Sun J, Sheng C, Wang Z, Wang Y, Zhang C, Fan R. Systematic review and meta-analysis of efficacy of mesenchymal stem cells on locomotor recovery in animal models of traumatic brain injury. Stem Cell Res Ther. 2015 Mar 26;6(1):47. doi: 10.1186/s13287-015-0034-0. PMID 25881229
- [Background] Pischiutta F, Caruso E, Lugo A, Cavaleiro H, Stocchetti N, Citerio G, Salgado A, Gallus S, Zanier ER. Systematic review and meta-analysis of preclinical studies testing mesenchymal stromal cells for traumatic brain injury. NPJ Regen Med. 2021 Oct 29;6(1):71. doi: 10.1038/s41536-021-00182-8. PMID 34716332
- [Background] Kabat M, Bobkov I, Kumar S, Grumet M. Trends in mesenchymal stem cell clinical trials 2004-2018: Is efficacy optimal in a narrow dose range? Stem Cells Transl Med. 2020 Jan;9(1):17-27. doi: 10.1002/sctm.19-0202. Epub 2019 Dec 5. PMID 31804767
- [Background] Wakabayashi K, Nagai A, Sheikh AM, Shiota Y, Narantuya D, Watanabe T, Masuda J, Kobayashi S, Kim SU, Yamaguchi S. Transplantation of human mesenchymal stem cells promotes functional improvement and increased expression of neurotrophic factors in a rat focal cerebral ischemia model. J Neurosci Res. 2010 Apr;88(5):1017-25. doi: 10.1002/jnr.22279. PMID 19885863
- [Background] Xu C, Fu F, Li X, Zhang S. Mesenchymal stem cells maintain the microenvironment of central nervous system by regulating the polarization of macrophages/microglia after traumatic brain injury. Int J Neurosci. 2017 Dec;127(12):1124-1135. doi: 10.1080/00207454.2017.1325884. Epub 2017 May 19. PMID 28464695
- [Background] Darkazalli A, Vied C, Badger CD, Levenson CW. Human Mesenchymal Stem Cell Treatment Normalizes Cortical Gene Expression after Traumatic Brain Injury. J Neurotrauma. 2017 Jan 1;34(1):204-212. doi: 10.1089/neu.2015.4322. Epub 2016 Jun 10. PMID 27161121
- [Background] Lazarus HM, Haynesworth SE, Gerson SL, Rosenthal NS, Caplan AI. Ex vivo expansion and subsequent infusion of human bone marrow-derived stromal progenitor cells (mesenchymal progenitor cells): implications for therapeutic use. Bone Marrow Transplant. 1995 Oct;16(4):557-64. PMID 8528172
- [Background] Rodriguez-Fuentes DE, Fernandez-Garza LE, Samia-Meza JA, Barrera-Barrera SA, Caplan AI, Barrera-Saldana HA. Mesenchymal Stem Cells Current Clinical Applications: A Systematic Review. Arch Med Res. 2021 Jan;52(1):93-101. doi: 10.1016/j.arcmed.2020.08.006. Epub 2020 Sep 22. PMID 32977984
- [Background] Zhuang WZ, Lin YH, Su LJ, Wu MS, Jeng HY, Chang HC, Huang YH, Ling TY. Mesenchymal stem/stromal cell-based therapy: mechanism, systemic safety and biodistribution for precision clinical applications. J Biomed Sci. 2021 Apr 14;28(1):28. doi: 10.1186/s12929-021-00725-7. PMID 33849537
- [Background] Thompson M, Mei SHJ, Wolfe D, Champagne J, Fergusson D, Stewart DJ, Sullivan KJ, Doxtator E, Lalu M, English SW, Granton J, Hutton B, Marshall J, Maybee A, Walley KR, Santos CD, Winston B, McIntyre L. Cell therapy with intravascular administration of mesenchymal stromal cells continues to appear safe: An updated systematic review and meta-analysis. EClinicalMedicine. 2020 Jan 17;19:100249. doi: 10.1016/j.eclinm.2019.100249. eCollection 2020 Feb. PMID 31989101
- [Background] Kawabori M, Weintraub AH, Imai H, Zinkevych I, McAllister P, Steinberg GK, Frishberg BM, Yasuhara T, Chen JW, Cramer SC, Achrol AS, Schwartz NE, Suenaga J, Lu DC, Semeniv I, Nakamura H, Kondziolka D, Chida D, Kaneko T, Karasawa Y, Paadre S, Nejadnik B, Bates D, Stonehouse AH, Richardson RM, Okonkwo DO. Cell Therapy for Chronic TBI: Interim Analysis of the Randomized Controlled STEMTRA Trial. Neurology. 2021 Feb 22;96(8):e1202-e1214. doi: 10.1212/WNL.0000000000011450. PMID 33397772
- [Background] Wang S, Cheng H, Dai G, Wang X, Hua R, Liu X, Wang P, Chen G, Yue W, An Y. Umbilical cord mesenchymal stem cell transplantation significantly improves neurological function in patients with sequelae of traumatic brain injury. Brain Res. 2013 Sep 26;1532:76-84. doi: 10.1016/j.brainres.2013.08.001. Epub 2013 Aug 11. PMID 23942181
- [Background] Tian C, Wang X, Wang X, Wang L, Wang X, Wu S, Wan Z. Autologous bone marrow mesenchymal stem cell therapy in the subacute stage of traumatic brain injury by lumbar puncture. Exp Clin Transplant. 2013 Apr;11(2):176-81. doi: 10.6002/ect.2012.0053. Epub 2012 Aug 11. PMID 22891928
- [Background] Zhang ZX, Guan LX, Zhang K, Zhang Q, Dai LJ. A combined procedure to deliver autologous mesenchymal stromal cells to patients with traumatic brain injury. Cytotherapy. 2008;10(2):134-9. doi: 10.1080/14653240701883061. PMID 18368592
- [Background] Vaquero J, Zurita M, Bonilla C, Fernandez C, Rubio JJ, Mucientes J, Rodriguez B, Blanco E, Donis L. Progressive increase in brain glucose metabolism after intrathecal administration of autologous mesenchymal stromal cells in patients with diffuse axonal injury. Cytotherapy. 2017 Jan;19(1):88-94. doi: 10.1016/j.jcyt.2016.10.001. Epub 2016 Nov 2. PMID 27816409
- [Background] Schepici G, Silvestro S, Bramanti P, Mazzon E. Traumatic Brain Injury and Stem Cells: An Overview of Clinical Trials, the Current Treatments and Future Therapeutic Approaches. Medicina (Kaunas). 2020 Mar 19;56(3):137. doi: 10.3390/medicina56030137. PMID 32204311
- [Background] Cox CS Jr, Baumgartner JE, Harting MT, Worth LL, Walker PA, Shah SK, Ewing-Cobbs L, Hasan KM, Day MC, Lee D, Jimenez F, Gee A. Autologous bone marrow mononuclear cell therapy for severe traumatic brain injury in children. Neurosurgery. 2011 Mar;68(3):588-600. doi: 10.1227/NEU.0b013e318207734c. PMID 21192274
- [Background] Liao GP, Harting MT, Hetz RA, Walker PA, Shah SK, Corkins CJ, Hughes TG, Jimenez F, Kosmach SC, Day MC, Tsao K, Lee DA, Worth LL, Baumgartner JE, Cox CS Jr. Autologous bone marrow mononuclear cells reduce therapeutic intensity for severe traumatic brain injury in children. Pediatr Crit Care Med. 2015 Mar;16(3):245-55. doi: 10.1097/PCC.0000000000000324. PMID 25581630
- [Background] Cox CS Jr, Hetz RA, Liao GP, Aertker BM, Ewing-Cobbs L, Juranek J, Savitz SI, Jackson ML, Romanowska-Pawliczek AM, Triolo F, Dash PK, Pedroza C, Lee DA, Worth L, Aisiku IP, Choi HA, Holcomb JB, Kitagawa RS. Treatment of Severe Adult Traumatic Brain Injury Using Bone Marrow Mononuclear Cells. Stem Cells. 2017 Apr;35(4):1065-1079. doi: 10.1002/stem.2538. Epub 2016 Nov 23. PMID 27800660
- [Background] Leibacher J, Henschler R. Biodistribution, migration and homing of systemically applied mesenchymal stem/stromal cells. Stem Cell Res Ther. 2016 Jan 11;7:7. doi: 10.1186/s13287-015-0271-2. PMID 26753925
- [Background] Armitage J, Tan DBA, Troedson R, Young P, Lam KV, Shaw K, Sturm M, Weiss DJ, Moodley YP. Mesenchymal stromal cell infusion modulates systemic immunological responses in stable COPD patients: a phase I pilot study. Eur Respir J. 2018 Mar 1;51(3):1702369. doi: 10.1183/13993003.02369-2017. Print 2018 Mar. No abstract available. PMID 29348155
- [Background] Matthay MA, Calfee CS, Zhuo H, Thompson BT, Wilson JG, Levitt JE, Rogers AJ, Gotts JE, Wiener-Kronish JP, Bajwa EK, Donahoe MP, McVerry BJ, Ortiz LA, Exline M, Christman JW, Abbott J, Delucchi KL, Caballero L, McMillan M, McKenna DH, Liu KD. Treatment with allogeneic mesenchymal stromal cells for moderate to severe acute respiratory distress syndrome (START study): a randomised phase 2a safety trial. Lancet Respir Med. 2019 Feb;7(2):154-162. doi: 10.1016/S2213-2600(18)30418-1. Epub 2018 Nov 16. PMID 30455077
- [Background] Zheng G, Huang L, Tong H, Shu Q, Hu Y, Ge M, Deng K, Zhang L, Zou B, Cheng B, Xu J. Treatment of acute respiratory distress syndrome with allogeneic adipose-derived mesenchymal stem cells: a randomized, placebo-controlled pilot study. Respir Res. 2014 Apr 4;15(1):39. doi: 10.1186/1465-9921-15-39. PMID 24708472
- [Background] Wilson JG, Liu KD, Zhuo H, Caballero L, McMillan M, Fang X, Cosgrove K, Vojnik R, Calfee CS, Lee JW, Rogers AJ, Levitt J, Wiener-Kronish J, Bajwa EK, Leavitt A, McKenna D, Thompson BT, Matthay MA. Mesenchymal stem (stromal) cells for treatment of ARDS: a phase 1 clinical trial. Lancet Respir Med. 2015 Jan;3(1):24-32. doi: 10.1016/S2213-2600(14)70291-7. Epub 2014 Dec 17. PMID 25529339
- [Background] Yip HK, Fang WF, Li YC, Lee FY, Lee CH, Pei SN, Ma MC, Chen KH, Sung PH, Lee MS. Human Umbilical Cord-Derived Mesenchymal Stem Cells for Acute Respiratory Distress Syndrome. Crit Care Med. 2020 May;48(5):e391-e399. doi: 10.1097/CCM.0000000000004285. PMID 32187077
- [Background] Simonson OE, Mougiakakos D, Heldring N, Bassi G, Johansson HJ, Dalen M, Jitschin R, Rodin S, Corbascio M, El Andaloussi S, Wiklander OP, Nordin JZ, Skog J, Romain C, Koestler T, Hellgren-Johansson L, Schiller P, Joachimsson PO, Hagglund H, Mattsson M, Lehtio J, Faridani OR, Sandberg R, Korsgren O, Krampera M, Weiss DJ, Grinnemo KH, Le Blanc K. In Vivo Effects of Mesenchymal Stromal Cells in Two Patients With Severe Acute Respiratory Distress Syndrome. Stem Cells Transl Med. 2015 Oct;4(10):1199-213. doi: 10.5966/sctm.2015-0021. Epub 2015 Aug 18. PMID 26285659
- [Background] Qu W, Wang Z, Hare JM, Bu G, Mallea JM, Pascual JM, Caplan AI, Kurtzberg J, Zubair AC, Kubrova E, Engelberg-Cook E, Nayfeh T, Shah VP, Hill JC, Wolf ME, Prokop LJ, Murad MH, Sanfilippo FP. Cell-based therapy to reduce mortality from COVID-19: Systematic review and meta-analysis of human studies on acute respiratory distress syndrome. Stem Cells Transl Med. 2020 Sep;9(9):1007-1022. doi: 10.1002/sctm.20-0146. Epub 2020 May 29. PMID 32472653
- [Background] Leng Z, Zhu R, Hou W, Feng Y, Yang Y, Han Q, Shan G, Meng F, Du D, Wang S, Fan J, Wang W, Deng L, Shi H, Li H, Hu Z, Zhang F, Gao J, Liu H, Li X, Zhao Y, Yin K, He X, Gao Z, Wang Y, Yang B, Jin R, Stambler I, Lim LW, Su H, Moskalev A, Cano A, Chakrabarti S, Min KJ, Ellison-Hughes G, Caruso C, Jin K, Zhao RC. Transplantation of ACE2- Mesenchymal Stem Cells Improves the Outcome of Patients with COVID-19 Pneumonia. Aging Dis. 2020 Mar 9;11(2):216-228. doi: 10.14336/AD.2020.0228. eCollection 2020 Apr. PMID 32257537
- [Background] Chen J, Hu C, Chen L, Tang L, Zhu Y, Xu X, Chen L, Gao H, Lu X, Yu L, Dai X, Xiang C, Li L. Clinical Study of Mesenchymal Stem Cell Treatment for Acute Respiratory Distress Syndrome Induced by Epidemic Influenza A (H7N9) Infection: A Hint for COVID-19 Treatment. Engineering (Beijing). 2020 Oct;6(10):1153-1161. doi: 10.1016/j.eng.2020.02.006. Epub 2020 Feb 28. PMID 32292627
- [Background] Chang Y, Park SH, Huh JW, Lim CM, Koh Y, Hong SB. Intratracheal administration of umbilical cord blood-derived mesenchymal stem cells in a patient with acute respiratory distress syndrome. J Korean Med Sci. 2014 Mar;29(3):438-40. doi: 10.3346/jkms.2014.29.3.438. Epub 2014 Feb 27. PMID 24616596
- [Background] Shi L, Huang H, Lu X, Yan X, Jiang X, Xu R, Wang S, Zhang C, Yuan X, Xu Z, Huang L, Fu JL, Li Y, Zhang Y, Yao WQ, Liu T, Song J, Sun L, Yang F, Zhang X, Zhang B, Shi M, Meng F, Song Y, Yu Y, Wen J, Li Q, Mao Q, Maeurer M, Zumla A, Yao C, Xie WF, Wang FS. Effect of human umbilical cord-derived mesenchymal stem cells on lung damage in severe COVID-19 patients: a randomized, double-blind, placebo-controlled phase 2 trial. Signal Transduct Target Ther. 2021 Feb 10;6(1):58. doi: 10.1038/s41392-021-00488-5. PMID 33568628
- [Background] Shu L, Niu C, Li R, Huang T, Wang Y, Huang M, Ji N, Zheng Y, Chen X, Shi L, Wu M, Deng K, Wei J, Wang X, Cao Y, Yan J, Feng G. Treatment of severe COVID-19 with human umbilical cord mesenchymal stem cells. Stem Cell Res Ther. 2020 Aug 18;11(1):361. doi: 10.1186/s13287-020-01875-5. PMID 32811531
- [Background] Adas G, Cukurova Z, Yasar KK, Yilmaz R, Isiksacan N, Kasapoglu P, Yesilbag Z, Koyuncu ID, Karaoz E. The Systematic Effect of Mesenchymal Stem Cell Therapy in Critical COVID-19 Patients: A Prospective Double Controlled Trial. Cell Transplant. 2021 Jan-Dec;30:9636897211024942. doi: 10.1177/09636897211024942. PMID 34180719
- [Background] Lanzoni G, Linetsky E, Correa D, Messinger Cayetano S, Alvarez RA, Kouroupis D, Alvarez Gil A, Poggioli R, Ruiz P, Marttos AC, Hirani K, Bell CA, Kusack H, Rafkin L, Baidal D, Pastewski A, Gawri K, Lenero C, Mantero AMA, Metalonis SW, Wang X, Roque L, Masters B, Kenyon NS, Ginzburg E, Xu X, Tan J, Caplan AI, Glassberg MK, Alejandro R, Ricordi C. Umbilical cord mesenchymal stem cells for COVID-19 acute respiratory distress syndrome: A double-blind, phase 1/2a, randomized controlled trial. Stem Cells Transl Med. 2021 May;10(5):660-673. doi: 10.1002/sctm.20-0472. Epub 2021 Jan 5. PMID 33400390
- [Background] Dilogo IH, Aditianingsih D, Sugiarto A, Burhan E, Damayanti T, Sitompul PA, Mariana N, Antarianto RD, Liem IK, Kispa T, Mujadid F, Novialdi N, Luviah E, Kurniawati T, Lubis AMT, Rahmatika D. Umbilical cord mesenchymal stromal cells as critical COVID-19 adjuvant therapy: A randomized controlled trial. Stem Cells Transl Med. 2021 Sep;10(9):1279-1287. doi: 10.1002/sctm.21-0046. Epub 2021 Jun 8. PMID 34102020
- [Background] Xu X, Jiang W, Chen L, Xu Z, Zhang Q, Zhu M, Ye P, Li H, Yu L, Zhou X, Zhou C, Chen X, Zheng X, Xu K, Cai H, Zheng S, Jiang W, Wu X, Li D, Chen L, Luo Q, Wang Y, Qu J, Li Y, Zheng W, Jiang Y, Tang L, Xiang C, Li L. Evaluation of the safety and efficacy of using human menstrual blood-derived mesenchymal stromal cells in treating severe and critically ill COVID-19 patients: An exploratory clinical trial. Clin Transl Med. 2021 Feb;11(2):e297. doi: 10.1002/ctm2.297. PMID 33634996
- [Background] Meng F, Xu R, Wang S, Xu Z, Zhang C, Li Y, Yang T, Shi L, Fu J, Jiang T, Huang L, Zhao P, Yuan X, Fan X, Zhang JY, Song J, Zhang D, Jiao Y, Liu L, Zhou C, Maeurer M, Zumla A, Shi M, Wang FS. Human umbilical cord-derived mesenchymal stem cell therapy in patients with COVID-19: a phase 1 clinical trial. Signal Transduct Target Ther. 2020 Aug 27;5(1):172. doi: 10.1038/s41392-020-00286-5. PMID 32855385
- [Background] Iglesias M, Butron P, Torre-Villalvazo I, Torre-Anaya EA, Sierra-Madero J, Rodriguez-Andoney JJ, Tovar-Palacio AR, Zentella-Dehesa A, Dominguez-Cherit G, Rodriguez-Reyna TS, Granados-Arriola J, Espisosa-Cruz V, Tellez-Pallares FP, Lozada-Estrada A, Zepeda Carrillo CA, Vazquez-Mezquita AJ, Nario-Chaidez HF. Mesenchymal Stem Cells for the Compassionate Treatment of Severe Acute Respiratory Distress Syndrome Due to COVID 19. Aging Dis. 2021 Apr 1;12(2):360-370. doi: 10.14336/AD.2020.1218. eCollection 2021 Apr. PMID 33815870
- [Background] Saleh M, Vaezi AA, Aliannejad R, Sohrabpour AA, Kiaei SZF, Shadnoush M, Siavashi V, Aghaghazvini L, Khoundabi B, Abdoli S, Chahardouli B, Seyhoun I, Alijani N, Verdi J. Cell therapy in patients with COVID-19 using Wharton's jelly mesenchymal stem cells: a phase 1 clinical trial. Stem Cell Res Ther. 2021 Jul 16;12(1):410. doi: 10.1186/s13287-021-02483-7. PMID 34271988
- [Background] Sanchez-Guijo F, Garcia-Arranz M, Lopez-Parra M, Monedero P, Mata-Martinez C, Santos A, Sagredo V, Alvarez-Avello JM, Guerrero JE, Perez-Calvo C, Sanchez-Hernandez MV, Del-Pozo JL, Andreu EJ, Fernandez-Santos ME, Soria-Juan B, Hernandez-Blasco LM, Andreu E, Sempere JM, Zapata AG, Moraleda JM, Soria B, Fernandez-Aviles F, Garcia-Olmo D, Prosper F. Adipose-derived mesenchymal stromal cells for the treatment of patients with severe SARS-CoV-2 pneumonia requiring mechanical ventilation. A proof of concept study. EClinicalMedicine. 2020 Aug;25:100454. doi: 10.1016/j.eclinm.2020.100454. Epub 2020 Jul 10. PMID 32838232
- [Background] Hashemian SR, Aliannejad R, Zarrabi M, Soleimani M, Vosough M, Hosseini SE, Hossieni H, Keshel SH, Naderpour Z, Hajizadeh-Saffar E, Shajareh E, Jamaati H, Soufi-Zomorrod M, Khavandgar N, Alemi H, Karimi A, Pak N, Rouzbahani NH, Nouri M, Sorouri M, Kashani L, Madani H, Aghdami N, Vasei M, Baharvand H. Mesenchymal stem cells derived from perinatal tissues for treatment of critically ill COVID-19-induced ARDS patients: a case series. Stem Cell Res Ther. 2021 Jan 29;12(1):91. doi: 10.1186/s13287-021-02165-4. PMID 33514427
- [Background] Liang B, Chen J, Li T, Wu H, Yang W, Li Y, Li J, Yu C, Nie F, Ma Z, Yang M, Xiao M, Nie P, Gao Y, Qian C, Hu M. Clinical remission of a critically ill COVID-19 patient treated by human umbilical cord mesenchymal stem cells: A case report. Medicine (Baltimore). 2020 Jul 31;99(31):e21429. doi: 10.1097/MD.0000000000021429. PMID 32756149
- [Background] Tang L, Jiang Y, Zhu M, Chen L, Zhou X, Zhou C, Ye P, Chen X, Wang B, Xu Z, Zhang Q, Xu X, Gao H, Wu X, Li D, Jiang W, Qu J, Xiang C, Li L. Clinical study using mesenchymal stem cells for the treatment of patients with severe COVID-19. Front Med. 2020 Oct;14(5):664-673. doi: 10.1007/s11684-020-0810-9. Epub 2020 Aug 6. PMID 32761491
- [Background] Nair AB, Jacob S. A simple practice guide for dose conversion between animals and human. J Basic Clin Pharm. 2016 Mar;7(2):27-31. doi: 10.4103/0976-0105.177703. PMID 27057123
- [Background] Czeiter E, Amrein K, Gravesteijn BY, Lecky F, Menon DK, Mondello S, Newcombe VFJ, Richter S, Steyerberg EW, Vyvere TV, Verheyden J, Xu H, Yang Z, Maas AIR, Wang KKW, Buki A; CENTER-TBI Participants and Investigators. Blood biomarkers on admission in acute traumatic brain injury: Relations to severity, CT findings and care path in the CENTER-TBI study. EBioMedicine. 2020 Jun;56:102785. doi: 10.1016/j.ebiom.2020.102785. Epub 2020 May 25. PMID 32464528
- [Background] Huie JR, Mondello S, Lindsell CJ, Antiga L, Yuh EL, Zanier ER, Masson S, Rosario BL, Ferguson AR; Transforming Research and Clinical Knowledge in Traumatic Brain Injury (TRACK-TBI) Investigators, The Transforming Research and Clinical Knowledge in Traumatic Brain Injury (TRACK-TBI) Investigators, Collaborative European NeuroTrauma Effectiveness Research in Traumatic Brain Injury (CENTER-TBI) Participants and Investigators, Collaborative European NeuroTrauma Effectiveness Research in Traumatic Brain Injury (CENTER-TBI) Participants and Investigators. Biomarkers for Traumatic Brain Injury: Data Standards and Statistical Considerations. J Neurotrauma. 2021 Sep 15;38(18):2514-2529. doi: 10.1089/neu.2019.6762. Epub 2020 Apr 1. PMID 32046588
- [Background] Maas AIR, Menon DK, Manley GT, Abrams M, Akerlund C, Andelic N, Aries M, Bashford T, Bell MJ, Bodien YG, Brett BL, Buki A, Chesnut RM, Citerio G, Clark D, Clasby B, Cooper DJ, Czeiter E, Czosnyka M, Dams-O'Connor K, De Keyser V, Diaz-Arrastia R, Ercole A, van Essen TA, Falvey E, Ferguson AR, Figaji A, Fitzgerald M, Foreman B, Gantner D, Gao G, Giacino J, Gravesteijn B, Guiza F, Gupta D, Gurnell M, Haagsma JA, Hammond FM, Hawryluk G, Hutchinson P, van der Jagt M, Jain S, Jain S, Jiang JY, Kent H, Kolias A, Kompanje EJO, Lecky F, Lingsma HF, Maegele M, Majdan M, Markowitz A, McCrea M, Meyfroidt G, Mikolic A, Mondello S, Mukherjee P, Nelson D, Nelson LD, Newcombe V, Okonkwo D, Oresic M, Peul W, Pisica D, Polinder S, Ponsford J, Puybasset L, Raj R, Robba C, Roe C, Rosand J, Schueler P, Sharp DJ, Smielewski P, Stein MB, von Steinbuchel N, Stewart W, Steyerberg EW, Stocchetti N, Temkin N, Tenovuo O, Theadom A, Thomas I, Espin AT, Turgeon AF, Unterberg A, Van Praag D, van Veen E, Verheyden J, Vyvere TV, Wang KKW, Wiegers EJA, Williams WH, Wilson L, Wisniewski SR, Younsi A, Yue JK, Yuh EL, Zeiler FA, Zeldovich M, Zemek R; InTBIR Participants and Investigators. Traumatic brain injury: progress and challenges in prevention, clinical care, and research. Lancet Neurol. 2022 Nov;21(11):1004-1060. doi: 10.1016/S1474-4422(22)00309-X. Epub 2022 Sep 29. PMID 36183712
- [Background] Marion CM, Radomski KL, Cramer NP, Galdzicki Z, Armstrong RC. Experimental Traumatic Brain Injury Identifies Distinct Early and Late Phase Axonal Conduction Deficits of White Matter Pathophysiology, and Reveals Intervening Recovery. J Neurosci. 2018 Oct 10;38(41):8723-8736. doi: 10.1523/JNEUROSCI.0819-18.2018. Epub 2018 Aug 24. PMID 30143572
- [Background] Hulkower MB, Poliak DB, Rosenbaum SB, Zimmerman ME, Lipton ML. A decade of DTI in traumatic brain injury: 10 years and 100 articles later. AJNR Am J Neuroradiol. 2013 Nov-Dec;34(11):2064-74. doi: 10.3174/ajnr.A3395. Epub 2013 Jan 10. PMID 23306011
- [Background] Lepinoux-Chambaud C, Eyer J. Review on intermediate filaments of the nervous system and their pathological alterations. Histochem Cell Biol. 2013 Jul;140(1):13-22. doi: 10.1007/s00418-013-1101-1. Epub 2013 Jun 8. PMID 23749407
- [Background] Shahim P, Zetterberg H, Tegner Y, Blennow K. Serum neurofilament light as a biomarker for mild traumatic brain injury in contact sports. Neurology. 2017 May 9;88(19):1788-1794. doi: 10.1212/WNL.0000000000003912. Epub 2017 Apr 12. PMID 28404801
- [Background] Hossain I, Mohammadian M, Takala RSK, Tenovuo O, Lagerstedt L, Ala-Seppala H, Frantzen J, van Gils M, Hutchinson P, Katila AJ, Maanpaa HR, Menon DK, Newcombe VF, Tallus J, Hrusovsky K, Wilson DH, Blennow K, Sanchez JC, Zetterberg H, Posti JP. Early Levels of Glial Fibrillary Acidic Protein and Neurofilament Light Protein in Predicting the Outcome of Mild Traumatic Brain Injury. J Neurotrauma. 2019 May 15;36(10):1551-1560. doi: 10.1089/neu.2018.5952. Epub 2019 Jan 8. PMID 30489229
- [Background] Zetterberg H, Hietala MA, Jonsson M, Andreasen N, Styrud E, Karlsson I, Edman A, Popa C, Rasulzada A, Wahlund LO, Mehta PD, Rosengren L, Blennow K, Wallin A. Neurochemical aftermath of amateur boxing. Arch Neurol. 2006 Sep;63(9):1277-80. doi: 10.1001/archneur.63.9.1277. PMID 16966505
- [Background] Shahim P, Gren M, Liman V, Andreasson U, Norgren N, Tegner Y, Mattsson N, Andreasen N, Ost M, Zetterberg H, Nellgard B, Blennow K. Serum neurofilament light protein predicts clinical outcome in traumatic brain injury. Sci Rep. 2016 Nov 7;6:36791. doi: 10.1038/srep36791. PMID 27819296
- [Background] Graham NSN, Zimmerman KA, Moro F, Heslegrave A, Maillard SA, Bernini A, Miroz JP, Donat CK, Lopez MY, Bourke N, Jolly AE, Mallas EJ, Soreq E, Wilson MH, Fatania G, Roi D, Patel MC, Garbero E, Nattino G, Baciu C, Fainardi E, Chieregato A, Gradisek P, Magnoni S, Oddo M, Zetterberg H, Bertolini G, Sharp DJ. Axonal marker neurofilament light predicts long-term outcomes and progressive neurodegeneration after traumatic brain injury. Sci Transl Med. 2021 Sep 29;13(613):eabg9922. doi: 10.1126/scitranslmed.abg9922. Epub 2021 Sep 29. PMID 34586833
- [Background] Shahim P, Politis A, van der Merwe A, Moore B, Chou YY, Pham DL, Butman JA, Diaz-Arrastia R, Gill JM, Brody DL, Zetterberg H, Blennow K, Chan L. Neurofilament light as a biomarker in traumatic brain injury. Neurology. 2020 Aug 11;95(6):e610-e622. doi: 10.1212/WNL.0000000000009983. Epub 2020 Jul 8. PMID 32641538
- [Background] Lange RT, Lippa S, Brickell TA, Gill J, French LM. Serum Tau, Neurofilament Light Chain, Glial Fibrillary Acidic Protein, and Ubiquitin Carboxyl-Terminal Hydrolase L1 Are Associated with the Chronic Deterioration of Neurobehavioral Symptoms after Traumatic Brain Injury. J Neurotrauma. 2023 Mar;40(5-6):482-492. doi: 10.1089/neu.2022.0249. Epub 2022 Oct 18. PMID 36170576
- [Background] Newcombe VFJ, Ashton NJ, Posti JP, Glocker B, Manktelow A, Chatfield DA, Winzeck S, Needham E, Correia MM, Williams GB, Simren J, Takala RSK, Katila AJ, Maanpaa HR, Tallus J, Frantzen J, Blennow K, Tenovuo O, Zetterberg H, Menon DK. Post-acute blood biomarkers and disease progression in traumatic brain injury. Brain. 2022 Jun 30;145(6):2064-2076. doi: 10.1093/brain/awac126. PMID 35377407
- [Background] Korley FK, Jain S, Sun X, Puccio AM, Yue JK, Gardner RC, Wang KKW, Okonkwo DO, Yuh EL, Mukherjee P, Nelson LD, Taylor SR, Markowitz AJ, Diaz-Arrastia R, Manley GT; TRACK-TBI Study Investigators. Prognostic value of day-of-injury plasma GFAP and UCH-L1 concentrations for predicting functional recovery after traumatic brain injury in patients from the US TRACK-TBI cohort: an observational cohort study. Lancet Neurol. 2022 Sep;21(9):803-813. doi: 10.1016/S1474-4422(22)00256-3. PMID 35963263
- [Background] Helmrich IRAR, Czeiter E, Amrein K, Buki A, Lingsma HF, Menon DK, Mondello S, Steyerberg EW, von Steinbuchel N, Wang KKW, Wilson L, Xu H, Yang Z, van Klaveren D, Maas AIR; CENTER-TBI participants and investigators. Incremental prognostic value of acute serum biomarkers for functional outcome after traumatic brain injury (CENTER-TBI): an observational cohort study. Lancet Neurol. 2022 Sep;21(9):792-802. doi: 10.1016/S1474-4422(22)00218-6. PMID 35963262
- [Background] Gardner RC, Rubenstein R, Wang KKW, Korley FK, Yue JK, Yuh EL, Mukherje P, Valadka AB, Okonkwo DO, Diaz-Arrastia R, Manley GT. Age-Related Differences in Diagnostic Accuracy of Plasma Glial Fibrillary Acidic Protein and Tau for Identifying Acute Intracranial Trauma on Computed Tomography: A TRACK-TBI Study. J Neurotrauma. 2018 Oct 15;35(20):2341-2350. doi: 10.1089/neu.2018.5694. Epub 2018 Jun 29. PMID 29717620
- [Background] Papa L, Silvestri S, Brophy GM, Giordano P, Falk JL, Braga CF, Tan CN, Ameli NJ, Demery JA, Dixit NK, Mendes ME, Hayes RL, Wang KK, Robertson CS. GFAP out-performs S100beta in detecting traumatic intracranial lesions on computed tomography in trauma patients with mild traumatic brain injury and those with extracranial lesions. J Neurotrauma. 2014 Nov 15;31(22):1815-22. doi: 10.1089/neu.2013.3245. Epub 2014 Sep 12. PMID 24903744
- [Background] Thelin EP, Zeiler FA, Ercole A, Mondello S, Buki A, Bellander BM, Helmy A, Menon DK, Nelson DW. Serial Sampling of Serum Protein Biomarkers for Monitoring Human Traumatic Brain Injury Dynamics: A Systematic Review. Front Neurol. 2017 Jul 3;8:300. doi: 10.3389/fneur.2017.00300. eCollection 2017. PMID 28717351
- [Background] Kuhle J, Gaiottino J, Leppert D, Petzold A, Bestwick JP, Malaspina A, Lu CH, Dobson R, Disanto G, Norgren N, Nissim A, Kappos L, Hurlbert J, Yong VW, Giovannoni G, Casha S. Serum neurofilament light chain is a biomarker of human spinal cord injury severity and outcome. J Neurol Neurosurg Psychiatry. 2015 Mar;86(3):273-9. doi: 10.1136/jnnp-2013-307454. Epub 2014 Jun 16. PMID 24935984
- [Background] Kuhle J, Kropshofer H, Haering DA, Kundu U, Meinert R, Barro C, Dahlke F, Tomic D, Leppert D, Kappos L. Blood neurofilament light chain as a biomarker of MS disease activity and treatment response. Neurology. 2019 Mar 5;92(10):e1007-e1015. doi: 10.1212/WNL.0000000000007032. Epub 2019 Feb 8. PMID 30737333
- [Background] Scott G, Zetterberg H, Jolly A, Cole JH, De Simoni S, Jenkins PO, Feeney C, Owen DR, Lingford-Hughes A, Howes O, Patel MC, Goldstone AP, Gunn RN, Blennow K, Matthews PM, Sharp DJ. Minocycline reduces chronic microglial activation after brain trauma but increases neurodegeneration. Brain. 2018 Feb 1;141(2):459-471. doi: 10.1093/brain/awx339. PMID 29272357
- [Background] Petrou P, Kassis I, Ginzberg A, Hallimi M, Karussis D. Effects of Mesenchymal Stem Cell Transplantation on Cerebrospinal Fluid Biomarkers in Progressive Multiple Sclerosis. Stem Cells Transl Med. 2022 Mar 3;11(1):55-58. doi: 10.1093/stcltm/szab017. PMID 35641166
- [Background] Husain M. Smarter adaptive platform clinical trials in neurology. Brain. 2022 Apr 18;145(2):409-410. doi: 10.1093/brain/awac005. No abstract available. PMID 35435950
- [Background] Gaipa G, Introna M, Golay J, Nolli ML, Vallanti G, Parati E, Giordano R, Romagnoli L, Melazzini M, Biondi A, Biagi E. Development of advanced therapies in Italy: Management models and sustainability in six Italian cell factories. Cytotherapy. 2016 Apr;18(4):481-6. doi: 10.1016/j.jcyt.2016.01.002. PMID 26971677
- [Background] Sammali E, Alia C, Vegliante G, Colombo V, Giordano N, Pischiutta F, Boncoraglio GB, Barilani M, Lazzari L, Caleo M, De Simoni MG, Gaipa G, Citerio G, Zanier ER. Intravenous infusion of human bone marrow mesenchymal stromal cells promotes functional recovery and neuroplasticity after ischemic stroke in mice. Sci Rep. 2017 Jul 31;7(1):6962. doi: 10.1038/s41598-017-07274-w. PMID 28761170
- [Background] Introna M, Lucchini G, Dander E, Galimberti S, Rovelli A, Balduzzi A, Longoni D, Pavan F, Masciocchi F, Algarotti A, Mico C, Grassi A, Deola S, Cavattoni I, Gaipa G, Belotti D, Perseghin P, Parma M, Pogliani E, Golay J, Pedrini O, Capelli C, Cortelazzo S, D'Amico G, Biondi A, Rambaldi A, Biagi E. Treatment of graft versus host disease with mesenchymal stromal cells: a phase I study on 40 adult and pediatric patients. Biol Blood Marrow Transplant. 2014 Mar;20(3):375-81. doi: 10.1016/j.bbmt.2013.11.033. Epub 2013 Dec 7. PMID 24321746
- [Background] Dander E, Lucchini G, Vinci P, Introna M, Masciocchi F, Perseghin P, Balduzzi A, Bonanomi S, Longoni D, Gaipa G, Belotti D, Parma M, Algarotti A, Capelli C, Golay J, Rovelli A, Rambaldi A, Biondi A, Biagi E, D'Amico G. Mesenchymal stromal cells for the treatment of graft-versus-host disease: understanding the in vivo biological effect through patient immune monitoring. Leukemia. 2012 Jul;26(7):1681-4. doi: 10.1038/leu.2011.384. Epub 2012 Jan 13. No abstract available. PMID 22289986
- [Background] Lucchini G, Dander E, Pavan F, Di Ceglie I, Balduzzi A, Perseghin P, Gaipa G, Algarotti A, Introna M, Rambaldi A, Rovelli A, Biondi A, Biagi E, D'Amico G. Mesenchymal stromal cells do not increase the risk of viral reactivation nor the severity of viral events in recipients of allogeneic stem cell transplantation. Stem Cells Int. 2012;2012:690236. doi: 10.1155/2012/690236. Epub 2012 May 30. PMID 22701127
- [Background] Liang X, Ding Y, Zhang Y, Tse HF, Lian Q. Paracrine mechanisms of mesenchymal stem cell-based therapy: current status and perspectives. Cell Transplant. 2014;23(9):1045-59. doi: 10.3727/096368913X667709. PMID 23676629
- [Background] Acosta SA, Tajiri N, Hoover J, Kaneko Y, Borlongan CV. Intravenous Bone Marrow Stem Cell Grafts Preferentially Migrate to Spleen and Abrogate Chronic Inflammation in Stroke. Stroke. 2015 Sep;46(9):2616-27. doi: 10.1161/STROKEAHA.115.009854. Epub 2015 Jul 28. PMID 26219646
- [Background] Matthay MA, Pati S, Lee JW. Concise Review: Mesenchymal Stem (Stromal) Cells: Biology and Preclinical Evidence for Therapeutic Potential for Organ Dysfunction Following Trauma or Sepsis. Stem Cells. 2017 Feb;35(2):316-324. doi: 10.1002/stem.2551. Epub 2017 Jan 19. PMID 27888550
- [Background] Steyerberg EW, Mushkudiani N, Perel P, Butcher I, Lu J, McHugh GS, Murray GD, Marmarou A, Roberts I, Habbema JD, Maas AI. Predicting outcome after traumatic brain injury: development and international validation of prognostic scores based on admission characteristics. PLoS Med. 2008 Aug 5;5(8):e165; discussion e165. doi: 10.1371/journal.pmed.0050165. PMID 18684008
- [Background] A'Hern RP. Sample size tables for exact single-stage phase II designs. Stat Med. 2001 Mar 30;20(6):859-66. doi: 10.1002/sim.721. PMID 11252008
- [Background] Simon R, Wittes RE, Ellenberg SS. Randomized phase II clinical trials. Cancer Treat Rep. 1985 Dec;69(12):1375-81. PMID 4075313
- [Background] George MJ, Prabhakara K, Toledano-Furman NE, Wang YW, Gill BS, Wade CE, Olson SD, Cox CS Jr. Clinical Cellular Therapeutics Accelerate Clot Formation. Stem Cells Transl Med. 2018 Oct;7(10):731-739. doi: 10.1002/sctm.18-0015. Epub 2018 Aug 1. PMID 30070065
- [Background] Jung JW, Kwon M, Choi JC, Shin JW, Park IW, Choi BW, Kim JY. Familial occurrence of pulmonary embolism after intravenous, adipose tissue-derived stem cell therapy. Yonsei Med J. 2013 Sep;54(5):1293-6. doi: 10.3349/ymj.2013.54.5.1293. PMID 23918585
- [Background] Wu Z, Zhang S, Zhou L, Cai J, Tan J, Gao X, Zeng Z, Li D. Thromboembolism Induced by Umbilical Cord Mesenchymal Stem Cell Infusion: A Report of Two Cases and Literature Review. Transplant Proc. 2017 Sep;49(7):1656-1658. doi: 10.1016/j.transproceed.2017.03.078. PMID 28838459
- [Background] Rubio D, Garcia-Castro J, Martin MC, de la Fuente R, Cigudosa JC, Lloyd AC, Bernad A. Spontaneous human adult stem cell transformation. Cancer Res. 2005 Apr 15;65(8):3035-9. doi: 10.1158/0008-5472.CAN-04-4194. PMID 15833829 (Retraction: PMID 20710046 de la Fuente R, Bernad A, Garcia-Castro J, Martin MC, Cigudosa JC. Cancer Res. 2010 Aug 15;70(16):6682)
- [Background] Rosland GV, Svendsen A, Torsvik A, Sobala E, McCormack E, Immervoll H, Mysliwietz J, Tonn JC, Goldbrunner R, Lonning PE, Bjerkvig R, Schichor C. Long-term cultures of bone marrow-derived human mesenchymal stem cells frequently undergo spontaneous malignant transformation. Cancer Res. 2009 Jul 1;69(13):5331-9. doi: 10.1158/0008-5472.CAN-08-4630. Epub 2009 Jun 9. PMID 19509230
- [Background] de la Fuente R, Bernad A, Garcia-Castro J, Martin MC, Cigudosa JC. Retraction: Spontaneous human adult stem cell transformation. Cancer Res. 2010 Aug 15;70(16):6682. doi: 10.1158/0008-5472.CAN-10-2451. No abstract available. PMID 20710046
- [Background] Torsvik A, Rosland GV, Svendsen A, Molven A, Immervoll H, McCormack E, Lonning PE, Primon M, Sobala E, Tonn JC, Goldbrunner R, Schichor C, Mysliwietz J, Lah TT, Motaln H, Knappskog S, Bjerkvig R. Spontaneous malignant transformation of human mesenchymal stem cells reflects cross-contamination: putting the research field on track - letter. Cancer Res. 2010 Aug 1;70(15):6393-6. doi: 10.1158/0008-5472.CAN-10-1305. Epub 2010 Jul 14. No abstract available. PMID 20631079
- [Background] Garcia S, Bernad A, Martin MC, Cigudosa JC, Garcia-Castro J, de la Fuente R. Pitfalls in spontaneous in vitro transformation of human mesenchymal stem cells. Exp Cell Res. 2010 May 15;316(9):1648-50. doi: 10.1016/j.yexcr.2010.02.016. Epub 2010 Feb 18. No abstract available. PMID 20171963
- [Background] Toyserkani NM, Jorgensen MG, Tabatabaeifar S, Jensen CH, Sheikh SP, Sorensen JA. Concise Review: A Safety Assessment of Adipose-Derived Cell Therapy in Clinical Trials: A Systematic Review of Reported Adverse Events. Stem Cells Transl Med. 2017 Sep;6(9):1786-1794. doi: 10.1002/sctm.17-0031. Epub 2017 Jul 19. PMID 28722289